CLINICAL TRIAL: NCT00217581
Title: Phase II Trial of Bevacizumab, Docetaxel, and Oxaliplatin in Gastric and Gastroesophageal Junction Cancer
Brief Title: Bevacizumab, Oxaliplatin, and Docetaxel in Treating Patients With Locally Advanced Unresectable or Metastatic Stomach or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Philip Philip, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441641; P30CA022453 (NIH); WSU-D-2840; UMCC-2005-052; AVENTIS-WSU-D-2840
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2014-07-07 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: recurrent gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Bevacizumab; Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel, Oxaliplatin & Bevacizumab (Experimental): Must be administered 1st before Docetaxel & Oxaliplatin.7.5 mg/kg, IV, day 1 of each cycle; During the first cycle, bevacizumab will be delivered over 90 + or - 15 minutes. If the 1st IV infusion is tolerated w/o infusion-associated adverse events, the 2nd infusion may be delivered over 60 + or - 10 minutes. If the 60 min infusion is well tolerated, all subsequent infusions may be delivered over 30 min + or - 10 mins.
  Interventions: Biological: Bevacizumab; Drug: Docetaxel; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Bevacizumab — Must be administered 1st before Docetaxel & Oxaliplatin.7.5 mg/kg, IV, day 1 of each cycle; During the first cycle, bevacizumab will be delivered over 90 + or - 15 minutes. If the 1st IV infusion is tolerated w/o infusion-associated adverse events, the 2nd infusion may be delivered over 60 + or - 10 minutes. If the 60 min infusion is well tolerated, all subsequent infusions may be delivered over 30 min + or - 10 mins.
  Other Names: Avastin
Drug: Docetaxel — Must be administered 2nd after Bevacizumab and followed by Oxaliplatin.70 mg/m(2), IV over 60 minutes, day 1 of each cycle;
  Other Names: Taxotere
Drug: Oxaliplatin — Must be administered 3rd after Bevacizumab and Docetaxel. 75 mg/m(2), IV over 120 minutes, Day 1 of each cycle.
  Other Names: Eloxatin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as oxaliplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with oxaliplatin and docetaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with oxaliplatin and docetaxel works in treating patients with locally advanced unresectable or metastatic stomach or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with locally advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma treated with bevacizumab, oxaliplatin, and docetaxel.

Secondary

* Determine the response rate in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine time to treatment failure and overall survival of patients treated with this regimen.
* Determine the changes in general and disease-specific quality of life, in terms of response to treatment, in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes, oxaliplatin IV over 120 minutes, and docetaxel IV over 60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses beyond CR.

After completion of study treatment, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 38 patients will be accrued for this study within 18-23 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric or gastroesophageal junction adenocarcinoma

  * Locally advanced unresectable or metastatic disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10mm by spiral CT scan

  * Bone metastases, ascites, or pleural effusions are not considered measurable disease
  * Evaluable disease must be present outside previously irradiated field
* No CNS or brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* SWOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 mg/dL
* No evidence of bleeding diathesis or coagulopathy

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ ULN
* INR < 1.5

Renal

* Creatinine < 2.0 mg/dL
* Urine protein:creatinine ratio < 1.0

Cardiovascular

* No history of deep venous thrombosis requiring anticoagulation
* No active angina
* No myocardial infarction within the past year
* No cerebrovascular accident within the past year
* No uncontrolled hypertension (systolic blood pressure [BP] > 170 mm Hg and/or diastolic BP > 100 mm Hg) despite medical management

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No peripheral neuropathy > grade 1
* No history of allergy to any of the study drugs or drugs formulated with polysorbate 80
* No known HIV infection
* No active peptic ulcer disease
* No serious non-healing wound, ulcer, or bone fracture
* No unresolved bacterial infection requiring antibiotics
* No other active malignancy within the past 3 years except for cancers that have been treated with a curative intent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy for gastric cancer unless disease relapsed > 6 months after completion of non-taxane adjuvant chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since radiotherapy

Surgery

* At least 4 weeks since prior surgery or open biopsy (except indwelling venous catheter placement)
* No concurrent surgery

Other

* At least 4 weeks since prior and no concurrent participation in another experimental drug trial
* No concurrent full-dose anticoagulation
* No concurrent experimental drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Principal Investigator — Barbara Ann Karmanos Cancer Institute; Basil El-Rayes, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (4):
- United States (4):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel, Oxaliplatin & Bevacizumab: Must be administered 1st before Docetaxel & Oxaliplatin.7.5 mg/kg, IV, day 1 of each cycle; During the first cycle, bevacizumab will be delivered over 90 + or - 15 minutes. If the 1st IV infusion is tolerated w/o infusion-associated adverse events, the 2nd infusion may be delivered over 60 + or - 10 minutes. If the 60 min infusion is well tolerated, all subsequent infusions may be delivered over 30 min + or - 10 mins.
  Bevacizumab: Must be administered 1st before Docetaxel & Oxaliplatin.7.5 mg/kg, IV, day 1 of each cycle; During the first cycle, bevacizumab will be delivered over 90 + or - 15 minutes. If the 1st IV infusion is tolerated w/o infusion-associated adverse events, the 2nd infusion may be delivered over 60 + or - 10 minutes.
Period: Overall Study
Arm/Group | Docetaxel, Oxaliplatin & Bevacizumab
Started | 39
Completed | 38
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel, Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: After every 2 cycles (1 cycle =21 days) From study registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel, Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 38
months | 6.6 [4.4 to 10.5]

2. Secondary Outcome: Response Rate by RECIST Criteria
Description: Percentage of Participants with response by RECIST criteria until progression
Time Frame: After every 2 cycles (1 cycle =21 days)
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Docetaxel, Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 38
percentage of responders | 42 [28 to 58]

3. Secondary Outcome: Toxicity Profile
Description: Toxicity profile of grade 3 and grade 4 events using the NCI-CTCAE Version 3.0 scale for toxicity grading.
Time Frame: At 21 days following completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel, Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 38
Participants
  Neutropenia | 13
  Leukopenia | 1
  GI Perforation | 3
  TE Fistula | 1
  Hypertension | 2
  Venous Thromboemblism | 1
  Neuropathy | 5
  Nausea | 4
  Vomiting | 2
  Diarrhea | 3
  Dehydration | 4
  Fever | 2
  Fatigue | 2
  Anorexia | 2

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure using the Kaplan-Meier method
Time Frame: Every 21 days From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel, Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 38
months | 4.5 [3.6 to 6.3]

5. Secondary Outcome: Overall Survival
Description: Overall survival using the Kaplan-Meier method
Time Frame: Patients will be followed for survival every three months after they are off study or until their disease progresses, for up to two years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel, Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 38
months | 11.1 [8.2 to 15.3]

ADVERSE EVENTS:
Groups:
- Docetaxel, Oxaliplatin & Bevacizumab: Administered 1st before Docetaxel & Oxaliplatin.7.5 mg/kg, IV, day 1 of each cycle; 1st cycle, bevacizumab will be delivered over 90 +/- 15 mins. If the 1st IV infusion is tolerated w/o infusion-associated adverse events, the 2nd infusion may be delivered over 60 +/- 10 mins. If the 60 min infusion is well tolerated, all subsequent infusions may be delivered over 30 min +/- 10 mins.
  Bevacizumab: Administered 1st before Docetaxel & Oxaliplatin.7.5 mg/kg, IV, day 1 of each cycle; During the first cycle, bevacizumab will be delivered over 90 +/- 15 mins. If the 1st IV infusion is tolerated w/o infusion-associated adverse events, the 2nd infusion may be delivered over 60 +/- 10 mins. If the 60 min infusion is well tolerated, all subsequent infusions may be delivered over 30 min +/- 10 mins.
  Docetaxel: Must be administered 2nd after Bevacizumab then Oxaliplatin.70 mg/m(2), IV over 60 minutes, day 1 of each cycle;
Arm/Group | Docetaxel, Oxaliplatin & Bevacizumab
Serious Adverse Events (participants affected / at risk) | 23/39
Other Adverse Events (participants affected / at risk) | 23/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel, Oxaliplatin & Bevacizumab (N=39)
Neutrophils (Investigations) | 13 (13)
Nausea (Gastrointestinal disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Late Dehydration (Gastrointestinal disorders) | 3 (3)
Gastrointestinal (GI) Perforation (not graded) (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Acute Neuropathy (Nervous system disorders) | 2 (2)
White Blood Count (WBC) (Investigations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel, Oxaliplatin & Bevacizumab (N=39)
Nausea (Gastrointestinal disorders) | 10 (10)
Late Diarrhea (Gastrointestinal disorders) | 12 (12)
Fatigue (General disorders) | 14 (14)
Vomiting (Gastrointestinal disorders) | 4 (4)
Acute Neuropathy (Nervous system disorders) | 9 (9)
Hypertension (Vascular disorders) | 5 (5)
WBC (Investigations) | 2 (2)
Hemoglobin (HGB) (Investigations) | 3 (3)
Chronic Neuropathy (Nervous system disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
The trial completed its planned accrual. There were no significant limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No